CLINICAL TRIAL: NCT01595347
Title: Olive Oil's Cream Effectiveness in Prevention of Pressure Ulcers in Immobilized Patients in Primary Care.A Cluster Randomized Clinical Trial.
Brief Title: Olive Oil's Cream Effectiveness in Prevention of Pressure Ulcers in Immobilized Patients in Primary Care
Acronym: PrevenUP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Francisco Javier Navarro Moya, Effectiveness and Research Unit Coordinator. Distrito Sanitario Málaga., Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DSM-SAS-2012-1
Record Dates: First submitted 2012-01-10; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-01

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Primary Prevention; Fatty Acids; Vegetable Fats; Olive oil; "Pressure Ulcer[prevention and control]"[Mesh]
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyper-oxigenated fatty acid (Active Comparator): Hyper-oxigenated fatty acid,Equisetum arvense, Hypericum perforatum
  Interventions: Drug: Hyper-oxigenated fatty acid
- Olive oil's Cream (Experimental): Cream with 60% extra virgin olive oil.
  Interventions: Other: Olive oil's cream

INTERVENTIONS:
Drug: Hyper-oxigenated fatty acid — Aplicación tópica de Mepentol (R) en zonas de riesgo de úlceras por presión (sacro, caderas y talones) 1 aplicación/24 horas
  Arms: Hyper-oxigenated fatty acid
Other: Olive oil's cream — Application Olive oil's cream to 60% in areas at risk of pressure ulcers (sacrum, hips and heels) 1 application / 24 hours
  Arms: Olive oil's Cream

SUMMARY:
Pressure ulcers (UPP) represent an important sanitary problem affecting mostly elderly immobilized persons, increasing the burden of care to professionals in the health system, as well as pharmaceutical spending. There are studies of the effectiveness of various products in the prevention of the UPP, most made in hospitals and using fundamentally composed based on oily hyperbecome oxygenated acids (AGHO).

There do not exist studies realized specifically with cream of olive oil.

AIMS:

Principal: To verify the efficiency of a new intervention of UPP's prevention in immobilized patients consisting in the application of cream of olive oil. Secondary: To evaluate the cost - efficiency of this new intervention opposite to AGHO's application.

To value the degree of satisfaction of the patient and his keeper with regard to the use of cream of olive oil.

METHODOLOGY DESIGN: clinical Test randomized with two parallel branches. AREA: Population consultant of the health centers in the province of Malaga. SUBJECTS OF STUDY: Patients immobilized at the risk of developing UPP. INTERVENTION: Administration of cream of olive oil to the group of intervention and AGHO's administration to the group control. Follow-up for one year. VARIABLES. Principal variable: UPP's appearance. Secondary: Demographic and clinical data, presence of technical supports, information of the caragiver and questionnaire of satisfaction. STATISTICAL ANALYSIS: Test. Exact of Fischer. Odds's calculation ratio. Shapiro-Wilk's test. Parametric test t- student or test U of Mann-Whitney. Reason of the increase cost efficiency (ICER). Logistic regression model multivariant.

ELIGIBILITY:
Inclusion criteria:

* Patients with nursing diagnosis "risk of impaired skin integrity. "To determine this risk assessment tool we will use as the Braden scale. We will include only patients immobilized with increased risk of pressure ulcers (score less than or equal to 16).
* Patients with malnutrition or suspected malnutrition. To determine this state as an instrument we will use Mini Nutritional Assessment Scale "MNA" (score 10 points or less)
* Over 18 years.

Exclusion criteria:

* Patients refusal to participate in the study.
* Moved (patient no habitual residence in the health center where they make the study).
* Patients with plans to be out of the study area during the monitoring year.
* Hospitalized during the uptake phase of the sample
* Patient-terminal.
* Patient with the presence of pressure ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Appearance grade II pressure ulcers | 48 months
  The primary outcome or result is the appearance of grade II pressure ulcers in patients under study during the 9 months follow up. This will be confirmed by observation of the areas where we did the intervention (sacrum, hips and heels).

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Lupiáñez-Pérez, Enfermera, Study Chair — Distrito Sanitario Málaga. Servicio Andaluz de Salud; Leovigildo Ginel-Mendoza, Medico, Principal Investigator — Distrito Sanitario Málaga. Servicio Andaluz de Salud; Francisco Javier Navarro-Moya, Enfermero, Principal Investigator — Distrito Sanitario Málaga. Servicio Andaluz de Salud; Francisco Javier Martín-Santos, Enfermero, Principal Investigator — Distrito Sanitario Málaga. Servicio Andaluz de Salud; Rafaela Sepúlveda-Guerra, Enfermera, Principal Investigator — Distrito Sanitario Málaga. Servicio Andaluz de Salud; Rosa Vázquez-Cerdeiros, Enfermera, Principal Investigator — Distrito Sanitario Málaga. Servicio Andaluz de Salud
Locations (1):
- Distrito Sanitario Málaga. Servicio Andaluz de Salud, Málaga, Málaga, Spain

REFERENCES:
- [Derived] Lupianez-Perez I, Morilla-Herrera JC, Kaknani-Uttumchandani S, Lupianez-Perez Y, Cuevas-Fernandez-Gallego M, Martin-Santos F, Caro-Bautista J, Morales-Asencio JM. A cost minimization analysis of olive oil vs. hyperoxygenated fatty acid treatment for the prevention of pressure ulcers in primary healthcare: A randomized controlled trial. Wound Repair Regen. 2017 Sep;25(5):846-851. doi: 10.1111/wrr.12586. Epub 2017 Nov 6. PMID 28922519
- [Derived] Lupianez-Perez I, Uttumchandani SK, Morilla-Herrera JC, Martin-Santos FJ, Fernandez-Gallego MC, Navarro-Moya FJ, Lupianez-Perez Y, Contreras-Fernandez E, Morales-Asencio JM. Topical olive oil is not inferior to hyperoxygenated fatty aids to prevent pressure ulcers in high-risk immobilised patients in home care. Results of a multicentre randomised triple-blind controlled non-inferiority trial. PLoS One. 2015 Apr 17;10(4):e0122238. doi: 10.1371/journal.pone.0122238. eCollection 2015. PMID 25886152
- [Derived] Lupianez-Perez I, Morilla-Herrera JC, Ginel-Mendoza L, Martin-Santos FJ, Navarro-Moya FJ, Sepulveda-Guerra RP, Vazquez-Cerdeiros R, Cuevas-Fernandez-Gallego M, Benitez-Serrano IM, Lupianez-Perez Y, Morales-Asencio JM. Effectiveness of olive oil for the prevention of pressure ulcers caused in immobilized patients within the scope of primary health care: study protocol for a randomized controlled trial. Trials. 2013 Oct 23;14:348. doi: 10.1186/1745-6215-14-348. PMID 24152576